CLINICAL TRIAL: NCT02489305
Title: A Prospective, Longitudinal, Observational Study to Evaluate Potential Predictors of Relapse in Subjects With Major Depressive Disorder Who Have Responded to Antidepressant Treatment
Brief Title: Study to Evaluate Potential Predictors of Relapse in Participants With Major Depressive Disorder (MDD)
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR105160; OBSERVEMDD0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Depression; Anti-Depressant; Observational
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Major Depressive Disorder: Participants with major depressive disorder who have responded to oral antidepressant treatment will be observed over time.

SUMMARY:
The purpose of this study is to identify if there are self-reported or objective measures related to mood parameters that can predict near-term relapse (within 1 month or at another identified time point before meeting the criteria for relapse) or early symptomatic changes indicative of relapse prodrome in major depressive disorder (MDD).

DETAILED DESCRIPTION:
This is a prospective, multicenter, longitudinal, single-cohort, observational study in participants with MDD who have responded to, and are continuing to respond to and receive, an oral antidepressant treatment regimen. The study will consist of 2 parts: a screening phase of up to 2 weeks, and an observational phase of variable duration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have met Diagnostic and Statistical Manual of Mental Disorders-5th edition (DSM-V) criteria for diagnosis of nonpsychotic MDD within the past 2 years (that is, the start of the most recent major depressive episode (MDE) must be less than or equal to 24 Months before screening), as confirmed using the MINI International Neuropsychiatric Interview (MINI - DSM-V). MDD must be recurrent, rather than a single episode
* During the most recent MDE, participant must have responded to, and must be continuing to receive and respond to, an oral antidepressant treatment regimen (given at an adequate dosage and duration based on the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire), within the past 3 months. A change in the oral antidepressant treatment regimen since the time of achieving response in the most recent episode will be allowed
* Participants must have a Montgomery Asberg Depression Rating Scale total score less than or equal to 14
* Participant must be willing and able to complete self-reported assessments via a study-specific smartphone, and must be willing to wear an wrist actigraphy device for the duration of the study

Exclusion Criteria:

* Participant has any of the following DSM-V psychiatric diagnoses: MDD with psychotic features (lifetime), bipolar disorder (including lifetime diagnosis), schizophrenia, or schizoaffective disorder
* Participant has a history of drug or alcohol use, with a severity of at least moderate or severe, according to DSM-V criteria, within 6 months before screening
* Participant is currently receiving or has received vagal nerve stimulation (VNS), electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS) or deep brain stimulation (DBS) for the most recent MDE
* Participant is currently receiving stimulants, anticonvulsants, or mood stabilizers for treatment of his or her MDD
* Participant is a woman who is pregnant, or planning to become pregnant, while enrolled in this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with major depressive disorder who have responded to an oral antidepressant regimen will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Near Term Relapse | Baseline up to end of study (8 Weeks)
  Relapse will be defined as any of the following: a) MADRS total score greater than or equal to 22 on at least two consecutive visits, with an interval of 1-2 weeks; b) Hospitalization for worsening of depression; c) Suicidal ideation with intent, or suicidal behavior and d) Other (investigator will be asked to describe). MADRS total score ranges from 0 to 60, Higher scores represents a more severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (25):
- United States (25):
  - Birmingham, Alabama
  - Glendale, California
  - Oceanside, California
  - San Diego, California
  - Sherman Oaks, California
  - Stanford, California
  - Hartford, Connecticut
  - Jacksonville, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Skokie, Illinois
  - Springfield, Illinois
  - Iowa City, Iowa
  - Wichita, Kansas
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Li QS, Galbraith D, Morrison RL, Trivedi MH, Drevets WC. Circulating microRNA associated with future relapse status in major depressive disorder. Front Psychiatry. 2022 Aug 17;13:937360. doi: 10.3389/fpsyt.2022.937360. eCollection 2022. PMID 36061300